CLINICAL TRIAL: NCT02371187
Title: Does Dapagliflozin Augment The Favorable Adaptation To Endurance Exercise Training?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Bell (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-5529H
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): The dose of Dapagliflozin will begin as one 5 mg tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two 5 mg tablets per day for the remainder of the study.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Matching placebo for Dapagliflozin 5 mg will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin tablets, 5 mg, one per day for the first 14 days, increase to two per day for 70 days.
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Placebo — Matching placebo for Dapagliflozin 5 mg, one per day for the first 14 days, increase to two per day for 70 days.
  Arms: Placebo

SUMMARY:
Exercise is frequently prescribed as a favorable lifestyle intervention to prevent/reverse type 2 diabetes. It is also prescribed in addition to concurrent pharmacological treatment, such as metformin. Recent data (animal and human) suggest that metformin may attenuate the favorable benefits of exercise training. In light of the physiological mechanism of Dapagliflozin (sodium-glucose co-transporter 2 (SGLT2) inhibition), one might speculate that rather than inhibit, it will augment the favorable adaptations to exercise training.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double blind, repeated measures study. 30 sedentary adults will be recruited for participation and randomly assigned to one of two 12-week treatments: 1) supervised endurance exercise training 4 days per week plus daily oral administration of Dapagliflozin; 2) supervised endurance exercise training 4 days per week plus daily oral administration of placebo. Prior to and following completion of the treatment the following dependent variables will be quantified: a) maximal aerobic capacity; b) substrate utilization during standardized low-moderate intensity exercise; c) skeletal muscle aerobic enzyme activity; d) body composition; and, e) oral glucose tolerance, fasting glucose and insulin resistance.

The dose of Dapagliflozin will begin as 5 mg/day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to 10 mg/day for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. No known Type 2 Diabetes.
3. Body mass index 25-45 kg/m^2
4. Sedentary (maximum of 2/week regularly scheduled activity sessions of < 20 minutes during the previous 2 years).
5. Completion of a screening visit consisting of medical history, physical examination, and 12-lead electrocardiogram and blood pressure assessment at rest and during incremental exercise to volitional exhaustion (Note: Subjects with abnormal screening values may be eligible if the results are not clinically significant, as judged by the investigator or medical monitor).
6. Agree to abide by the study schedule and to return for the required assessments.
7. Be willing and able to repeatedly perform exercise.
8. Women of childbearing potential must have negative pregnancy test and be using acceptable contraception.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Evidence of clinically significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, hematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study or the safety of the subject, as judged by the investigator in agreement with the sponsor or medical monitor, have been hospitalized in the past 2 years as a result of these conditions, or are receiving pharmacological treatment for these conditions.
2. Use of prescription drugs (see exceptions listed below) or herbal preparations in the 4 weeks before study commencement.

   Permitted Prescription Drugs
   * Birth Control
   * Less than 7 days, short course antibiotics. Note: Rifampin is not permitted.
   * Other medicines, for gastroesophageal reflux disease (GERD), depression, seasonal allergies and over-the-counter analgesics, may be allowed, but will be approved on a case-by-case basis.
3. Is currently enrolled in another clinical study for another investigational drug or has taken any other investigational drug within 30 days before the screening visit.
4. Habitual and/or recent use (within 2 years) of tobacco.
5. Being considered unsuitable for participation in this trial for any reason, as judged by the investigator or medical monitor.
6. History of serious hypersensitivity reaction to Dapagliflozin.
7. Severe renal impairment, end-stage renal disease, or dialysis.
8. Pregnant or breastfeeding patients.
9. Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal and/or alanine aminotransferase (ALT) >3x upper limit of normal.
10. Total bilirubin >2.0 mg/dL (34.2 umol/L).
11. Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody Immunoglobulin M, Hepatitis B surface antigen and Hepatitis C virus antibody.
12. Estimated Glomerular Filtration Rate <60 mL/min/1.73 m^2 (calculated by Cockcroft-Gault formula).
13. History of bladder cancer.
14. Recent cardiovascular events in a patient, including any of the following: acute coronary syndrome within 2 months prior to enrollment; hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment; acute stroke or trans-ischemic attack within two months prior to enrollment; less than two months post coronary artery re-vascularization; congestive heart failure defined as New York Heart Association class IV, unstable or acute congestive heart failure. Note: eligible patients with congestive heart failure,especially those who are on diuretic therapy, should have careful monitoring of their volume status throughout the study.
15. Blood pressure at enrollment: Systolic blood pressure ≥165 mmHg and/or diastolic blood pressure ≥100 mmHg.
16. Blood pressure at randomization: Systolic blood pressure ≥165 mmHg and/or diastolic blood pressure ≥100 mmHg
17. Patients who, in the judgment of the medical monitor, may be at risk for dehydration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newman AA, Grimm NC, Wilburn JR, Schoenberg HM, Trikha SRJ, Luckasen GJ, Biela LM, Melby CL, Bell C. Influence of Sodium Glucose Cotransporter 2 Inhibition on Physiological Adaptation to Endurance Exercise Training. J Clin Endocrinol Metab. 2019 Jun 1;104(6):1953-1966. doi: 10.1210/jc.2018-01741. PMID 30597042

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 18 | 19
Completed | 15 | 15
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: Participants who were withdrawn for various reasons were excluded from the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 30
Height [Mean (Standard Deviation); unit: meters] | 1.67 (0.08) | 1.71 (0.10) | 1.69 (8.92)
Body Mass [Mean (Standard Deviation); unit: Kilograms] | 87.8 (17.3) | 91.8 (16.9) | 89.80 (16.9)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meters squared] | 31.3 (5.4) | 31.2 (4.3) | 31.3 (4.77)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeter of mercury] | 130 (14) | 129 (13) | 129.5 (13)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 83 (10) | 82 (11) | 83 (10.5)
Peak Oxygen Uptake [Mean (Standard Deviation); unit: milliliter per kilogram per minute] | 26.9 (5.3) | 30.1 (6.1) | 27.49 (5.7)
Fasting Glucose [Mean (Standard Deviation); unit: milligrams per deciliter] | 78.8 (7.3) | 75.8 (5.1) | 77.3 (5.9)
Fasting Insulin [Mean (Standard Deviation); unit: MilliUnits per Liter] | 7.6 (4.0) | 8.9 (6.7) | 8.3 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Maximal Oxygen Uptake at Week 12
Description: Indirect calorimetry
Time Frame: Baseline,12 weeks
Measure: Mean (Standard Deviation); unit: Milliliters/Kilogram/Minute
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 15 | 15
Milliliters/Kilogram/Minute
  Pre-Exercise Training | 26.9 (5.3) | 30.1 (6.1)
  Post-Exercise Training | 30.6 (6.1) | 32.4 (7.5)

2. Primary Outcome: Change From Baseline of Respiratory Exchange Ratio at Week 12
Description: The respiratory exchange ratio (RER) is the ratio between the amount of carbon dioxide (CO2) produced in metabolism and oxygen (O2) used during standardized exercise.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: Respiratory Exchange Ratio
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 15 | 15
Respiratory Exchange Ratio
  Pre-Exercise Training | 1.91 (0.05) | 1.16 (0.12)
  Post-Exercise Training | 1.19 (0.05) | 1.13 (0.06)

3. Primary Outcome: Change From Baseline of Maximal Aerobic Enzyme Activities in Skeletal Muscle at Week 12
Description: Maximal citrate synthase activity in skeletal muscle sample
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: micromol/min/miligram protein
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 15 | 15
micromol/min/miligram protein
  Pre-Exercise Training | 6.3 (3.7) | 5.8 (3.6)
  Post Exercise Training | 8.1 (4.5) | 8.0 (4.0)

4. Primary Outcome: Change From Baseline of Insulin Sensitivity at Week 12
Description: Insulin Sensitivity was estimated by measuring circulating glucose and insulin concentrations after a 12-hour fast and after ingestion of 75 g of glucose. Glucose was measured 5, 10, 15, 20, 30, 45, 60, 75, 90, 105 and 120 minutes after glucose ingestion. Insulin was measured 15, 30, 45, 60, 90 and 120 minutes after glucose ingestion. Insulin sensitivity was estimated using the Matsuda Index, represented by the formula: Matsuda index = 10,000/SQRT [fasting glucose*fasting insulin* (mean glucose from time 5, 10, 15, 20, 30, 45, 60, 75, 90, 105 and 120 minutes) * (mean insulin from time 15, 30, 45, 60, 90 and 120 minutes)], with higher numbers indicating better insulin sensitivity.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: MATSUDA Index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 15 | 15
MATSUDA Index
  Pre-Training | 8.7 (4.8) | 8.3 (4.9)
  Post-Training | 9.5 (4.8) | 12.9 (8.9)

5. Primary Outcome: Change From Baseline of Fat Free Mass at Week 12
Description: Via dual energy X-ray absorptiometry
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 15 | 15
Kilograms
  Pre-Exercise Training | 52 (9.9) | 57.8 (12.2)
  Post-Exercise Training | 52.2 (9.9) | 58.3 (12.1)

ADVERSE EVENTS:
Time Frame: Throughout the 12 week intervention period
Description: Subjects withdrawn are not included in the analysis of Baseline Characteristics and Outcome Measures, but are included for Adverse Events.
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 17/18 | 18/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=18) | Placebo (N=19)
Headaches and Dizziness (General disorders) | 4 (5) | 7 (7)
Cold Symptoms (General disorders) | 7 (8) | 10 (15)
Chest Congestion (General disorders) | 1 (1) | 2 (2)
General Stomach Pain and Diarrhea (General disorders) | 7 (7) | 5 (9)
Muscle soreness and joint pain (General disorders) | 8 (10) | 7 (9)
Urinary Disorders and Yeast Infections (General disorders) | 3 (3) | 3 (4)
Fatigue (General disorders) | 1 (1) | 1 (1)
Rash or skin irritation (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT02371187/Prot_SAP_ICF_000.pdf